CLINICAL TRIAL: NCT02550587
Title: Satisfaction Rate of Patients Receiving Anesthesia in the First Half of 2015, in Erzincan
Brief Title: Patient Satisfaction With Anesthesia Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cukurova University (Other)
Collaborators: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, Anaesthesiology and reanimation, Cukurova University
Other Study IDs: Erzincan Mengücek Gazi
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Anesthesia
Keywords: Patient Satisfaction; anesthesia Care
MeSH Terms: conditions — Patient Satisfaction | interventions — Physician Engagement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: satisfaction — anesthesia satisfaction rates

SUMMARY:
The level of patient satisfaction is an important indicator of health care quality because it causes to reconsider the functioning of the hospital and go to the new regulations. Postoperative thought gives us important information for improving the quality of anesthesia care and health care quality. The investigators aimed to investigate the status of the anesthesia satisfaction in patients.

DETAILED DESCRIPTION:
Patients will answer the questionnaire consisting of 15 questions

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing anesthesia
* between 18 - 65 years old
* to agree to participate in research
* undergo elective surgery

Exclusion Criteria:

* be a psychiatric disorder
* cardiovascular surgery
* Emergency surgery
* patients with speech-hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing anesthesia in Erzincan
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
anesthesia satisfaction rates | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Üniversity, Erzincan, Turkey (Türkiye)

REFERENCES:
- [Background] Fung D, Cohen MM. Measuring patient satisfaction with anesthesia care: a review of current methodology. Anesth Analg. 1998 Nov;87(5):1089-98. doi: 10.1097/00000539-199811000-00020. No abstract available. PMID 9806687
- [Background] Eberhart LH, Morin AM, Wulf H, Geldner G. Patient preferences for immediate postoperative recovery. Br J Anaesth. 2002 Nov;89(5):760-1. PMID 12393775
- [Background] Jenkins K, Grady D, Wong J, Correa R, Armanious S, Chung F. Post-operative recovery: day surgery patients' preferences. Br J Anaesth. 2001 Feb;86(2):272-4. doi: 10.1093/bja/86.2.272. PMID 11573673
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Mathur SK, Dube SK, Jain S. Knowledge about Anaesthesia and Anaesthesiologist Amongst General Population in India. Indian J Anaesth. 2009 Apr;53(2):179-86. PMID 20640120
- [Result] Demir A, Turan S, Balaban F, Karadeniz Ü, Erdemli Ö. Anestezi Uygulamaları ile İlgili Olarak Preanestezik Değerlendirme Sırasında Hastalarda Yapılan Anket Çalışması. Türk Anest Der Dergisi 2009;37:225-33